CLINICAL TRIAL: NCT02876289
Title: Retrospective Evaluation of Perampanel in a French Neurology and Epileptology Department (Hospices Civil de Lyon)
Acronym: PERLYON
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0556
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients treated with Perampanel
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel

SUMMARY:
Perampanel is a non-competitive antagonist of the AMPA ( 2-amino-3-(5-méthyl-3-hydroxy-1,2-oxazol-4-yl)) propanoïc acid receptors which was approved by the European Medicines Agency as adjunctive treatment for partial-onset seizures in patients 12 years and older, in 2012. The aim of this study is to evaluate effectiveness and safety of perampanel as add-on treatment in patients with refractory epilepsy.

The investigators retrospectively collected and analyzed the data of patients with refractory epilepsy who had been treated with perampanel between May of 2014 and April of 2015. In total, one hundred and ten patients were included (mean age 41 [SD = 15.2]). The mean duration of epilepsy was 25 years (SD = 14.4). The mean perampanel dose was 5.7 mg/d (SD = 2.3). The retention rate was 77% at 6 months and 61% at 12 months. After 6 months, the responder rate was 35.5%. Eight patients (7.3%) became seizure free. Adverse effects were reported in 60 patients (54.5%). Most common side effects were behaviour disturbance (22.7%), dizziness (15.5%), asthenia (11.8), somnolence (10%) and ataxia (9.1).

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory focal epilepsy
* Initiation of perampanel between 05/2014 and 04/2015

Exclusion Criteria:

* Exact date of initiation of Perampanel not defined
* Patients without follow-up data

Ages: 16 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with refractory focal epilepsy in which Perampanel were introduced between May 2014 and April 2015
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Retention rate | 6 months
  Proportion of patient still treated with Perampanel 6 months after its initiation

SECONDARY OUTCOMES:
Retention rate | 12 months
  Proportion of patients still treated with Perampanel 12 months after its initiation
Seizure freedom | 6 months
  Proportion of seizure-free patients during at least 6 months
Responder rates | 6 months
  Responder rates is defined as a reduction in seizure frequency of 50% or more compared with the three months before the initiation of perampanel.
Responder rates | 12 months
  Responder rates is defined as a reduction in seizure frequency of 50% or more compared with the three months before the initiation of perampanel.
Total withdrawal rate | 6 months
  Discontinuation rates at 6 months due to inefficiency or adverse effects
Total withdrawal rate | 12 months
  Discontinuation rates at 12 months due to inefficiency or adverse effects
Observed adverse effects during the observation period | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital neurologique, Lyon, France

IPD SHARING:
Plan to Share IPD: No